CLINICAL TRIAL: NCT02405975
Title: A Randomized Controlled Trial Assessing the Impact of an Online Educational Tool on Doctors' Knowledge and Confidence With Regards to Prescribing for Older Patients
Brief Title: RCT Assessing the Impact of Online Training on Doctors' Prescribing for Older Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Shane Cullinan, Research Pharmacist, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UCC-CUH-001
Record Dates: First submitted 2015-03-28; First posted 2015-04-01 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Appropriateness of Prescribing in Older Patients

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): These participants will not receive the educational intervention
- Intervention (Experimental): These participants will receive the online educational intervention "SCRIPT"
  Interventions: Other: SCRIPT

INTERVENTIONS:
Other: SCRIPT — An online tool designed to train doctors in all areas of prescribing
  Arms: Intervention

SUMMARY:
This study will assess, by means of a randomized controlled trial, the impact of an online educational tool, on doctors' knowledge and confidence with regards to prescribing for older patients.

DETAILED DESCRIPTION:
Both control and intervention groups will complete assessments at baseline, 4 weeks post intervention and 8 weeks post intervention.

Differences in mean test scores will be the primary outcome measure.

Qualitative information exploring doctors' attitudes and confidence, pre and post intervention will also be collected and will be a secondary outcome

ELIGIBILITY:
Inclusion Criteria:

* Registered non-consultant hospital doctor working in one of the hospitals approved by the ethics board

Exclusion Criteria:

* Currently working as a consultant
* Having previously worked as a pharmacist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Difference in mean test scores | At baseline, 4 weeks post intervention and 8 weeks post intervention
  test scores pre and post intervention compared

SECONDARY OUTCOMES:
Doctors' confidence with regards to prescribing for older patients | At baseline, 4 weeks post intervention and 8 weeks post intervention
  doctors answer a questionnaire as part of each assessment to determine their overall confidence with regards to prescribing for older patients

CONTACTS AND LOCATIONS:
Overall Officials: Shane Cullinan, BPharm, Principal Investigator — University College Cork
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland

REFERENCES:
- [Derived] Cullinan S, O'Mahony D, Byrne S. Use of an e-Learning Educational Module to Better Equip Doctors to Prescribe for Older Patients: A Randomised Controlled Trial. Drugs Aging. 2017 May;34(5):367-374. doi: 10.1007/s40266-017-0451-0. PMID 28258537